CLINICAL TRIAL: NCT05733416
Title: Intensive Cancer Screening After Cryptogenic Stroke (INCOGNITO) Pilot Randomized Trial
Brief Title: Intensive Cancer Screening After Cryptogenic Stroke
Acronym: INCOGNITO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Brain Canada (Other); Heart and Stroke Foundation of Canada (Other); Canadian Stroke Consortium (CSC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20230006-01H
Record Dates: First submitted 2023-01-28; First posted 2023-02-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Occult Cancer
Keywords: cryptogenic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Cancer Screening (Experimental): Usual care plus FDG PET/CT
  Interventions: Diagnostic Test: FDG PET/CT
- Usual Care (Other): Cancer screening according to sex, age and risk as per Canadian Task Force on Preventative Health Care)
  Interventions: Diagnostic Test: Usual Care

INTERVENTIONS:
Diagnostic Test: FDG PET/CT — F-fluorodeoxyglucose positron emission/computed tomography
  Arms: Intensive Cancer Screening
Diagnostic Test: Usual Care — Cancer screening according to sex, age and risk as per Canadian Task Force on Preventative Health Care
  Arms: Usual Care

SUMMARY:
The INCOGNITO Pilot Trial is a single centre pilot prospective randomized open-label blinded endpoint (PROBE) trial to assess the feasibility of a full-scale randomized trial to determine whether an occult cancer screening strategy of FDG PET/CT (F-fluorodeoxyglucose positron emission/computed tomography) in addition to usual care increases the number of occult cancers diagnosed after screening compared to usual care cancer screening alone in patients with cryptogenic stroke.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years
* presenting to the Ottawa Hospital Stroke Prevention Clinic or the Ottawa Hospital Neurovascular Unit with a first cryptogenic ischemic stroke after advanced evaluation as per American Heart Association guidelines and Saver approach (maximum 3 months after stroke)
* patient or delegate willing and able to provide informed consent.

Exclusion Criteria:

* contraindications to FDG PET/CT (pregnancy or unable to lie still in bed for 20 minutes)
* active cancer or previous cancer diagnosis (other than basal or squamous cell carcinoma of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment | Over 12 months
  Number of participants recruited

SECONDARY OUTCOMES:
Eligibility Rate | Over 12 months
  percentage of screened patients who are eligible
Consent Rate | Over 12 months
  percentage of eligible patients who provide consent
Retention Rate | Over 24 months
  percentage of participants retained at follow-up
Study Completion Rate | Over 24 months
  percentage of participants who completed all study procedures
Adherence Rate | Over 24 months
  adherence to screening strategy

OTHER OUTCOMES:
Screening time frame | Over 24 months
  time from diagnosis to screening
Reasons for participation | Over 24 months
  Reasons for accepting/declining participation
Usual care cancer screening strategies | Over 24 months
  Usual care cancer screening strategies ordered by treating physicians

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Dowlatshahi, MD PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No